CLINICAL TRIAL: NCT02282176
Title: A Randomised, Placebo Controlled Trial of Azithromycin for the Prevention of Chronic Lung Disease of Prematurity in Preterm Infants
Brief Title: TINN2: Treat Infection in NeoNates 2
Acronym: TINN2
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: University of Liverpool (Other); Cardiff University (Other); University of Nottingham (Other); Erasmus Medical Center (Other); Heinrich-Heine-Universität Düsseldorf (UDUS) (Unknown); Assistance Publique - Hôpitaux de Paris (Other); Mario Negri Institute (IRFMN) (Unknown); Advanced Biological Laboratories ABL (ABL SA) (Unknown); Simcyp Limited (SimCyp) (Unknown); Only For Children Pharmaceuticals (Industry); University of Ulm (Other); Karolinska Institutet (Other); Centre Hospitalier Chrétien (CHC) (Unknown); Semmelweis University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C12-75; 2013-003889-14 (EudraCT Number)
Record Dates: First submitted 2014-10-17; First posted 2014-11-04 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Neonates; Preterm; Azithromycin; Ureaplasma; Chronic Lung disease; Bronchopulmonary dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth | interventions — Azithromycin; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azithromycin (Experimental): 10mg/kg azithromycin IV daily (administered over a period of at least one 1 hour) for a period of 10 days.
  Interventions: Drug: Azithromycin
- Placebo (Placebo Comparator): Placebo IV daily (administered over a period of at least one 1 hour) for a period of 10 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — Azithromycin IV 10mg/kg daily for 10 days
  Arms: Azithromycin
Drug: Placebo — Azithromycin placebo (5% Dextrose) daily for 10 days
  Other Names: 5% Dextrose
  Arms: Placebo

SUMMARY:
The aim of the TINN2 study is to evaluate the efficacy of azithromycin in prevention of bronchopulmonary dysplasia in preterm neonates.

DETAILED DESCRIPTION:
In contrast to the situation in adults, most medicines used to treat the children of Europe have not been tested and are not authorised for use in children. In particular, 46% medicines prescribed to children in hospital are either unlicensed for their age group or, if licensed, are prescribed off label. Of the children who receive at least one medication in hospital, 67% receive an unlicensed or off-label drug, and in the context of intensive care, this rises to up to 90% of patients.

The new Paediatric Regulation entered into force in early 2007 ensure that medicines for use in children are of high quality, ethically evaluated and authorised appropriately. The Paediatric-Use Marketing Authorisation (PUMA) is a new type of marketing authorisation for drugs not covered by a patent, already available on the market for adults. PUMA applies to medicines lacking information and/or appropriate formulation for children of all ages.

Thus, the European Medicines Agency (EMA) has published a list of drugs, which azithromycin belongs, as priority medicinal products needing an evaluation in the paediatric population.

Bronchopulmonary dysplasia (BPD) is a specific disease of prematurity accompanied by pulmonary inflammation. Multiple factors may contribute to the occurrence of BPD. In infants who are at risk of developing CLD, one frequent finding is colonisation of the preterm lung with the microbe Ureaplasma.

Two Meta-Analyses and recent studies have suggested an association between the presence of pulmonary Ureaplasma and the development of BPD.

Azithromycin is a macrolide antibiotic active against Ureaplasma spp with anti-inflammatory properties. Thus, it may be effective in reducing the severity of bronchopulmonary diseases in which both infection and inflammation play a role.

TINN2 project: the aim of the TINN2 study is to evaluate the efficacy of azithromycin in prevention of bronchopulmonary dysplasia in preterm neonates. TINN2 is a consortium involving European leaders in neonatology, paediatric pharmacology, methodology and several SMEs that will establish links with ethical bodies and regulatory authorities.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-term, 28w + 6d gestational age (i.e. 28 weeks and 6 days, including infants born as one of a multiple birth)
2. Requirement for respiratory support within 12hrs of birth (intubated, or by noninvasive mechanical ventilation including continuous positive airway pressure)
3. Presence of an indwelling intravenous line for drug administration
4. Inborn, or born at site within the recruiting centre's neonatal network where follow up will be possible

Exclusion Criteria:

1. In the opinion of the PI, babies unlikely to survive until 48 hours after birth
2. Exposure to another macrolide antibiotic
3. Presence of major surgical or congenital abnormalities (not including patent ductus arteriosus or patent foramen ovale)
4. Infants born as part of a multiple pregnancy of three or more (i.e. triplets or more)
5. Contraindication of azithromycin as specified in the summary of characteristics of the product.
6. Participation in other clinical trials involving Investigational Medicinal Products (IMPs)

Ages: 23 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2017-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of surviving infants without CLD (Chronic Lung Disease) in the azithromycin treatment group when compared to placebo at 36 weeks post-menstrual age. | 36 weeks post-menstrual age

SECONDARY OUTCOMES:
Mortality rate (at 28 days, 36 weeks PMA, 2 years) | 28 days, 36 weeks PMA, 2 years
Severity of CLD (Chronic Lung Disease) according to NIH definition | 36 weeks PMA
Microbiology assessment | Baseline and days 5, 10, 21
  Microbiology assessment at baseline and days 5, 10, 21:
  Pulmonary colonisation by Ureaplasma spp. and Mycoplasma spp. (respiratory culture of endotracheal/nasopharyngeal aspirates and nasogastric aspirates (nasogastric only for Ureaplasma spp. at baseline) and species-specific quantitative PCR)
Inflammation Markers | Baseline and days 5, 10, 21
  Subroup of patients:
  Inflammatory markers at baseline and days 5, 10, 21 in plasma and bronchoalveolar lavage
  Identification of the following: IL-1, IL-6, IL-8, TNF-a, MCP-1, PMN/Am/TCC, C5a.
Duration of positive pressure respiratory support (i.e. conventional mechanical ventilation, nasal ventilation, continuous positive airway pressure, CPAP) and supplemental oxygen | up to 36 weeks PMA
Emergence of resistance to azithromycin in Ureaplasma spp. isolated from endotracheal or nasopharyngeal samples at baseline, days 5, 10 and 21 | Baseline, days 5, 10 and 21
  On each positive PCR a culture will be performed. Then, an antibiotic susceptibility testing upon positive cultures
Resistance to azithromycin among microbes isolated from stool or rectal swab obtained at baseline and day 21 | Baseline and day 21
  Antibiotic susceptibility testing on any identified microbes
Plasma concentrations | days 1, 3, 6 as required
  Each patients to be allocated two sample timepoints from the following schedule:
  Sample1:
  1 sample within 5 min after the end of dose administration (day 1) Or 1 sample at 6 hours after start of infusion (day 1) Or 1 sample at 12 hours after start of infusion (day 1)
  Sample 2:
  1 sample at 48 hours - just prior to the third administration (day 3) Or 1 sample at 144 hours- just prior to the sixth administration (day 6)
Exposure to antibiotics other than azithromycin during the hospital stay | up to 36weeks PMA
Development of complications of prematurity | 24 months
  Development of complications of prematurity: Nosocomial infection (sepsis, meningitis, pneumonia); intraventricular haemorrhage; necrotising enterocolitis; retinopathy of prematurity; patent ductus arteriosus; pulmonary hemorrhage, pneumothorax and pulmonary interstitial emphysema during hospital stay
Number of Adverse Events | 24 months
Number of participants with dysrhythmic episodes and QTc interval | 24 months
C-Reactive Protein | 24 months
Neurodevelopmental assessment: Assessment of neurodevelopment using the 3rd edition of the Bayley Scales of Infant Development at the corrected age of 24 months | 24 months
  Long-term follow up at the corrected age of 24 months
Respiratory function assessment: Assessment of respiratory symptoms using a validated International Study of Asthma and Allergies in Childhood (ISAAC) questionnaire | 24 months
  Long-term follow up at the corrected age of 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sailesh Kotecha, Principal Investigator — Cardiff University
Locations (16):
- Centre Hospitalier Chrétien (CHC), Liège, Belgium
- France (4):
  - Assistance Publique Hôpitaux de Paris (APHP), Paris
  - Inserm-Transfert (IT), Paris
  - Institut National de la Santé et de la Recherche Médicale (INSERM), Paris
  - Only for children pharmaceuticals (04CP), Paris
- Germany (2):
  - Heinrich-Heine-Universität Düsseldorf (UDUS), Düsseldorf
  - University of Ulm (UUlm), Ulm
- Hungary (2):
  - Semmelweis University Budapest, Faculty of Medicine (SOTE), Budapest
  - Pandy Kalman County Hospital, Gyula
- Mario Negri Institute (IRFMN), Milan, Italy
- Advanced Biological Laboratories ABL (ABL SA), Luxembourg, Luxembourg
- Erasmus-University Medical Center (ERAMUS), Rotterdam, Netherlands
- Karolinska Institutet (KI), Stockholm, Sweden
- United Kingdom (3):
  - Cardiff University (CU), Cardiff
  - University of Liverpool (UOL), Liverpool
  - Simcyp Limited (SimCyp), Sheffield

REFERENCES:
- [Background] Turner MA, Jacqz-Aigrain E, Kotecha S. Azithromycin, Ureaplasma and chronic lung disease of prematurity: a case study for neonatal drug development. Arch Dis Child. 2012 Jun;97(6):573-7. doi: 10.1136/adc.2010.195180. Epub 2011 Jun 22. PMID 21697219
- [Background] Pansieri C, Pandolfini C, Elie V, Turner MA, Kotecha S, Jacqz-Aigrain E, Bonati M. Ureaplasma, bronchopulmonary dysplasia, and azithromycin in European neonatal intensive care units: a survey. Sci Rep. 2014 Feb 12;4:4076. doi: 10.1038/srep04076. PMID 24518104
- [Background] Lowe J, Watkins WJ, Edwards MO, Spiller OB, Jacqz-Aigrain E, Kotecha SJ, Kotecha S. Association between pulmonary ureaplasma colonization and bronchopulmonary dysplasia in preterm infants: updated systematic review and meta-analysis. Pediatr Infect Dis J. 2014 Jul;33(7):697-702. doi: 10.1097/INF.0000000000000239. PMID 24445836
- See also: TINN2 website — http://tinn2-project.org/